CLINICAL TRIAL: NCT05744908
Title: Retrospective Evaluation of the Effectiveness of Oral Pentosan Polysulfate Treatment in the Improvement of Chronic Interstitial Cystitis Symptoms
Brief Title: Pentosan Polysulfate Treatment's Effectiveness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hisar Intercontinental Hospital (Other)
Responsible Party: Principal Investigator, Basri Cakiroglu, Principal Investigator, Hisar Intercontinental Hospital
Allocation: Randomized | Model: Sequential | Masking: Single | Purpose: Treatment
Other Study IDs: 10.01.2023/37
Record Dates: First submitted 2023-01-10; First posted 2023-02-27 (Actual); Last update posted 2025-05-22 (Actual); Status verified 2023-02

CONDITIONS: Chronic Interstitial Cystitis
MeSH Terms: conditions — Cystitis, Interstitial | interventions — Pentosan Sulfuric Polyester

STUDY DESIGN:
Intervention Model Description: two models: with and without Hunner's ulcer
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- With Hunner's ulcer (Active Comparator): Pentosan Polysulfate 100 mg
  Interventions: Other: Pentosan Polysulphate
- Without Hunner's ulcer (Active Comparator): Pentosan Polysulfate 100 mg
  Interventions: Other: Pentosan Polysulphate

INTERVENTIONS:
Other: Pentosan Polysulphate — 300mg 3 times a day

SUMMARY:
To examine the relationship between symptoms and quality of life before and after oral pentosan polysulfate (PPS) treatment in cases diagnosed with interstitial cystitis/painful bladder syndrome (IC/BPS).

DETAILED DESCRIPTION:
Demographic characteristics, medical history, clinical conditions, and laboratory and cystoscopic data of patients who applied to our clinic between January 2018 and December 2021 and were diagnosed with IC/BPS were retrospectively analyzed. Adult male and female patients with IC/BPS who received 300 mg/day PPS at least six months ago with complaints of pain, urge, frequency, and nocturia not associated with urinary tract infection were included in the study. In addition, pre- and post-treatment symptoms, ICSI scores, quality of life (scored between 1-4), and satisfaction were compared.

ELIGIBILITY:
Inclusion Criteria:

* Chronic interstitial cystitis
* Bladder Pain Syndrome

Exclusion Criteria:

* Acute cystitis
* Bladder cancer
* Chronic prostatitis
* Bladder stone
* Stress incontinence

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 37 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2023-01-10 (Actual)

PRIMARY OUTCOMES:
bladder wall thickness | Three months
  0.3 over 3 mm 1 under 3 mm,
improvement of lower urinary tract symptoms | Three months
  1 if symptoms improved, 0 if not

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Basri Cakiroglu, Istanbul
  - Hisar Intercontinental Hospital, Istanbul

IPD SHARING:
Plan to Share IPD: No